CLINICAL TRIAL: NCT06326164
Title: Effect of Kinesio-taping of Lower Limbs on Gait and Balance in Children With Diplegic Cerebral Palsy
Brief Title: Effect of Kinesio-taping of Lower Limbs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Khalil Sadeek, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sample
Record Dates: First submitted 2024-02-29; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy- Diplegia- Kinesio-taping- Balance- Gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Control group.
  Interventions: Procedure: kinesio-taping.
- Group B (Active Comparator): Experimental group.
  Interventions: Procedure: kinesio-taping.; Procedure: A designed physiotherapy program.

INTERVENTIONS:
Procedure: kinesio-taping. — A therapeutic tape that's applied strategically to the body to provide support, reduce pain, swelling and improve performance. Kinesio taping will be applied on both lower limbs. Taping will be applied for 4 days, 24 hours a day, on the lower limbs, and it will be removed for only one day per week.
Procedure: A designed physiotherapy program. — The designed physiotherapy program included passive stretching, weight bearing, muscle strengthening, functional exercises, neurodevelopmental treatment, splinting, balance training, and gait training. The treatment protocol will be repeated each session per weeks for twelve weeks.
  Arms: Group B

SUMMARY:
The goal of this clinical trail is to test if kinesio-taping on lower limbs has an effect on balance and gait in children with diplegic cerebral palsy. Children in study group will have designed physiotherapy for gait and balance, the control group will have designed physiotherapy in addition to kinesio-taping on both lower limbs.

DETAILED DESCRIPTION:
Diplegic cerebral palsy is the most prevalent type of cerebral palsy. The main challenge for spastic cerebral palsy is gross motor dysfunction. The motor problems of spastic cerebral palsy arise fundamentally from central nervous system dysfunction, which interferes in the development of normal alignment postural control against gravity and impedes normal motor development.

Positive effects of kinesio taping for improving range of motion in patients with different disorders are reported in some of the studies. In the present study, kinesio taping along with physiotherapy treatment is considered an effective method for postural control improvement in diplegic cerebral palsy children.

Given the importance of motion and functional mobility in daily life, design and execution of accurate scientific interventions is necessary for health care systems economically and ethically.

Research on this field and accurate analysis of functional mobility, spasticity, and range of motion are rare. The main goal of physical therapy in the rehabilitation of cerebral palsy is to improve motor function and increase the ability to control movement. therefore, the present study aims to explore the effects of kinesio taping of lower limbs on gait and balance of children with spastic diplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. A medical diagnosis of spastic diplegic cerebral palsy made by pediatricians or pediatric neurologists.
2. Children with spasticity grades ranged from 1 to 1 plus according to Modified ashworth scale.
3. Their age range from 6 to 10 years.
4. Children who can stand with poor balance and recognize and follow verbal orders and commands included in both testing and training techniques
5. No orthopedic surgeries

Exclusion Criteria:

1. Children who have skin sensitivity for using kinesio-taping.
2. A history of cardiac or orthopedic disability.
3. Children having visual or auditory defects.
4. They had a permanent deformity.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-18 (Estimated)

PRIMARY OUTCOMES:
Change in gait. | Change from Baseline gait at twelve weeks.
  Measurement of gait using Kinovea software.
Change in balance. | Change from Baseline balance at twelve weeks.
  Measurement of balance using the Biodex balance system.

CONTACTS AND LOCATIONS:
Overall Officials: A M KH, Bachelor's, Principal Investigator — Faculty of Physical Therapy Kafrelsheikh University; M B I, Ass. Prof, Study Chair — Faculty of physical therapy Kafrelsheikh university; O A AE, Professor, Study Chair — Faculty of medicine Kafrelshiekh university; S Y AE, lecturer, Study Director — Faculty of physical therapy Kafrelshiekh university
Locations (1):
- Asmaa Mohamed Khalil Sedeek, Kafr ash Shaykh, Egypt